CLINICAL TRIAL: NCT05674240
Title: Intrathecal Targeted Drug Delivery for Cancer Associated Pain
Brief Title: Prospective Evaluation of Intrathecal Targeted Drug Delivery for Cancer Associated Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00104840
Record Dates: First submitted 2022-12-14; First posted 2023-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer Pain; Chronic Pain; Cancer Associated Pain; Neuropathic Pain
Keywords: targeted drug delivery; cancer pain; conservative pain management; neuromodulation; opioid; healthcare-utilization; quality of life
MeSH Terms: conditions — Cancer Pain; Chronic Pain; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cancer associated pain treated with conservative medical management (CMM) only: Subjects in this group are patients who opted for conservative medical management for their chronic pain that is cancer associated, including physical therapy, oral or transdermal medications and injections
  Interventions: Combination Product: Conservative medical management
- Cancer associated pain treated with Intrathecal Drug Delivery system (IDDs) along with CMM: Patients in this group are those that opted for targeted drug delivery along with conservative medical management of their cancer-associated pain
  Interventions: Device: Intrathecal Targeted Drug Delivery; Combination Product: Conservative medical management

INTERVENTIONS:
Device: Intrathecal Targeted Drug Delivery — Intrathecal drug delivery systems (IDDs) deliver small doses of analgesics directly to the spinal cord.
  Other Names: Medtronic SynchroMed™ II pump
  Groups: Cancer associated pain treated with Intrathecal Drug Delivery system (IDDs) along with CMM
Combination Product: Conservative medical management — Including physical therapy, oral or transdermal medications and injections

SUMMARY:
This Registry study will prospectively evaluate the differences in treatment outcomes in terms of pain intensity, pain interference, concomitant medication use, health-related quality of life, opioid adverse effects, and healthcare utilization between targeted drug delivery and conservative medication management only groups.

DETAILED DESCRIPTION:
This is a prospective, open-label, short term patient registry where up to 169 subjects with cancer associated pain will be enrolled. Subjects with cancer associated pain who are receiving conservative medical management (CMM) only and cancer patients receiving Intrathecal Drug Delivery system (IDDs) along with CMM will be followed for up to 3 months. Subjects will be evaluated monthly up to 3 months from the medical care initiation which is the implant day for the IDDs group and start of the new treatment plan for the CMM group. Subjects that decide to cross-over to the IDDs group in a future date, will still be followed for their progress.

Based on routine care, subjects will be seen at day of implant, 1 month post-implant, 2 months post-implant, and 3- and 6- months post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 and older
* Uncontrolled cancer-associated pain (pain score of >5 on NRS) despite oral use of 60 mg/d morphine equivalent a week prior to screening
* Adverse side effects from long term opioid use defined as limiting or severely affecting patient's day to day function
* Life expectancy of > 3 months

Exclusion Criteria:

* Active infections
* Controlled pain without adverse side effects that are limiting day to day function
* Mechanical barriers
* Obstruction of Cerebrospinal Fluid (CSF)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 169 subjects with cancer-associated pain who are going to be treated either with conservative medical management (CMM) only or with Intrathecal Drug Delivery along with CMM per treatment plan.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity from Screening through 3-Months | 3-Months
  Change from baseline to Month 3 post treatment plan implementation in average pain as measured through Numerical Rating Scale (0-10 where higher scores mean worse outcome)
Change in Pain Interference from Screening through 3-Months | 3-Months
  Change from baseline to Month 3 post treatment plan implementation in pain interference as measured through Patient-Reported Outcomes Measurement Information System (PROMIS-29)

SECONDARY OUTCOMES:
Change in Drug Adverse Levels | 3-Months
  Average change from baseline to 3-Months in drug adverse levels as assessed through the Common Toxicity Criteria
Change in Oral Opioid Intake | 3-Months
  Average change from baseline to 3-Months in oral opioid intake
Change in Healthcare Utilization | 3-Months
  Average change from baseline to 3-Months in healthcare utilization as assessed by number of emergency, inpatient, and outpatient visits due to pain
Change in Patient Well-Being | 3-Months
  Average change from baseline to 3-Months in patient well-being as measured through Functional Assessment of Cancer Therapy: General (FACT-G) (0-4 where higher scores mean worse outcome)
Change in Patient Global Impression Change | 3-Months
  Average change from baseline to 3-Months in Patient Global Impression of Change (PGIC) (1-7 where higher scores mean better outcome)

OTHER OUTCOMES:
Change in Pain Intensity | 2-Months
  Change from baseline to 2-Months post treatment plan implementation in average pain as measured through Numerical Rating Scale (0-10 where higher scores mean worse outcome)
Change in Pain Interference | 2-Months
  Change from baseline to 2-Months post treatment plan implementation in pain interference as measured through Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Change in Drug Adverse Levels | 2-Months
  Average change from baseline to 2-Months in drug adverse levels as assessed through the Common Toxicity Criteria
Change in Oral Opioid Intake | 2-Months
  Average change from baseline to 2-Months in oral opioid intake
Change in Patient Well-Being | 2-Months
  Average change from baseline to 2-Months in patient well-being as measured through Functional Assessment of Cancer Therapy: General (FACT-G) (0-4 where higher scores mean worse outcome)
Change in Patient Global Impression Change | 2-Months
  Average change from baseline to 2-Months in Patient Global Impression of Change (PGIC) (1-7 where higher scores mean better outcome)
Change in Pain Intensity | 1-Month
  Change from baseline to 1-Month post treatment plan implementation in average pain as measured through Numerical Rating Scale (0-10 where higher scores mean worse outcome)
Change in Pain Interference | 1-Month
  Change from baseline to 1-Month post treatment plan implementation in pain interference as measured through Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Change in Drug Adverse Levels | 1-Month
  Average change from baseline to 1-Month in drug adverse levels as assessed through the Common Toxicity Criteria
Change in Oral Opioid Intake | 1-Month
  Average change from baseline to 1-Month in oral opioid intake
Change in Patient Well-Being | 1-Month
  Average change from baseline to 1-Month in patient well-being as measured through Functional Assessment of Cancer Therapy: General (FACT-G) (0-4 where higher scores mean worse outcome)
Change in Patient Global Impression Change | 1-Month
  Average change from baseline to 1-Month in Patient Global Impression of Change (PGIC) (1-7 where higher scores mean better outcome)
Average change from baseline to 6-Months in drug adverse levels as assessed through the Common Toxicity Criteria (NCI) | 6-Months
Average change from baseline to 6-Months in oral opioid intake | 6-Months
Average change from baseline to 6-Months in healthcare utilization as assessed by number of emergency, inpatient, and outpatient visits due to pain and length of hospital stays | 6-Months
Average change from baseline to 6-Months in patient well being as measured through FACT-G questionnaire | 6-Months
Overall patient satisfaction in 6-Months as assessed through PGIC questionnaire | 6-Months

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Littlefield, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Aurora Health, Oshkosh, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided